CLINICAL TRIAL: NCT07348718
Title: Rubix LS DKD Equity Registry (RUBIX-DKD): A Prospective Observational Patient Registry to Characterize Diabetic Kidney Disease Trajectories, Treatment Patterns, and Outcomes in Underserved Communities and to Enable a Future Embedded Phase IV Pragmatic Study
Brief Title: Rubix LS Diabetic Kidney Disease (DKD) Registry Study
Status: Active, not recruiting | Type: Observational
Sponsor: Rubix LS (Industry)
Responsible Party: Sponsor
Other Study IDs: RLS-DKD-REG-001
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: Diabetic Kidney Disease; Chronic Kidney Disease; Type 2 Diabetes Mellitus; Albuminuria; UACR; eGFR; CKD Progression; eGFR Slope; Patient Registry; Observational Study; Real-World Evidence; Health Equity; Social Determinants of Health; SGLT2 Inhibitor; Finerenone
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Albuminuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Kidney-Protective Therapies Used in Routine Care — Observed medication exposure during usual care (not assigned by the study), including ACE inhibitor/ARB therapy, SGLT2 inhibitors, nonsteroidal mineralocorticoid receptor antagonists, GLP-1 receptor agonists, and other clinician-directed therapies; exposure ascertained from the medical record.

SUMMARY:
Diabetic kidney disease (DKD) is a common complication of type 2 diabetes that can lead to kidney failure and increases the risk of cardiovascular disease. This prospective, observational patient registry will follow adults with type 2 diabetes and DKD who are receiving routine clinical care at participating sites, with intentional enrollment from underserved communities. Health information will be collected from medical records and brief questionnaires (including social and access factors) for up to 24 months to understand DKD progression, real-world treatment patterns, and outcomes. This study does not assign any treatment. With participant consent and appropriate privacy safeguards, de-identified registry data may be shared with researchers to accelerate evidence generation and inform future studies focused on improving outcomes.

DETAILED DESCRIPTION:
This study is a prospective, multi-site observational patient registry designed to characterize real-world diabetic kidney disease (DKD) trajectories, care patterns, and outcomes in care settings that serve underserved communities. The registry is intended to generate representative evidence that reflects routine clinical practice and to identify clinical and non-clinical factors that influence DKD progression and care delivery.

Participants will continue to receive all medical care as determined by their treating clinicians; no treatments, diagnostic tests, or clinical management decisions are assigned by the registry. Longitudinal data will be captured primarily from existing sources (e.g., electronic health records and, where available, linked administrative/claims data), including kidney function and albuminuria measures, cardiometabolic risk factors, comorbid conditions, medication exposure and persistence, clinically relevant safety events, and healthcare utilization. Participants will also be invited to complete brief questionnaires to capture patient-reported outcomes and social determinants of health (SDOH), including access and care barriers that may affect treatment initiation, monitoring, and outcomes.

The registry will support descriptive and comparative effectiveness analyses using appropriate observational methods to address confounding and missingness, and will enable development and validation of risk stratification and treatment-response models to inform precision therapy targeting and equitable implementation in real-world settings. A core emphasis is the creation of a high-quality, standardized dataset with clear provenance and data quality checks to support reproducible research.

Data sharing is a foundational component of the registry. With explicit participant consent and privacy safeguards, de-identified participant-level data and supporting documentation may be made available to qualified researchers under the data access approach described in the IPD sharing plan. Finally, findings and infrastructure developed through this registry (e.g., trial-ready sites, validated phenotypes, and risk models) are intended to inform the design of a subsequent Phase IV pragmatic study, which would be conducted under a separate protocol and separately registered, with re-contact and re-consent as applicable.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years at the time of enrollment

Documented diagnosis of type 2 diabetes mellitus in the medical record

Evidence of chronic kidney disease consistent with diabetic kidney disease (DKD), defined by one or more of the following, with evidence of chronicity (present for ≥3 months based on prior laboratory results, diagnosis codes, or clinician documentation):

eGFR <60 mL/min/1.73 m², and/or

Urine albumin-to-creatinine ratio (UACR) ≥30 mg/g

Receiving ongoing clinical care at a participating site with medical record data available for longitudinal follow-up

Able and willing to provide written informed consent (and authorization for medical record review, as applicable) and to complete registry questionnaires

Exclusion Criteria:

End-stage kidney disease at baseline (maintenance dialysis) or history of kidney transplant

Type 1 diabetes mellitus

Known primary kidney disease not primarily attributable to diabetes that, in the investigator's judgment, is expected to drive kidney outcomes (e.g., polycystic kidney disease, active glomerulonephritis, lupus nephritis, vasculitis)

Inability to provide informed consent or comply with registry procedures (e.g., no feasible longitudinal follow-up through the participating site)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with type 2 diabetes and chronic kidney disease consistent with diabetic kidney disease (e.g., reduced eGFR and/or elevated UACR) receiving routine clinical care at participating sites. Sites will primarily include safety-net systems, community hospitals, and FQHC-affiliated networks, with intentional enrollment strategies to ensure meaningful representation of underserved populations disproportionately affected by DKD. Longitudinal clinical data will be obtained from medical records, supplemented by participant questionnaires capturing patient-reported outcomes and social determinants of health.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Estimated Glomerular Filtration Rate (eGFR) Slope | 24 months
  Annualized change in kidney function, defined as the slope of estimated glomerular filtration rate (eGFR; mL/min/1.73m2/year) from baseline through 24 months. All available eGFR values obtained in routine clinical care during follow-up will be used. eGFR slope will be estimated using models that account for repeated measures (e.g., linear mixed-effects with random intercept/slope). Baseline eGFR is the value closest to enrollment; more negative slopes indicate faster decline.

SECONDARY OUTCOMES:
Time to DKD Progression Composite Outcome | 24 months
  Time from enrollment (baseline) to first occurrence of a DKD progression event, defined as any of the following: sustained ≥40% decline in eGFR from baseline confirmed by a repeat value ≥4 weeks apart; initiation of maintenance dialysis; kidney transplant; or kidney failure-related death. Events will be identified from routine clinical data (EHR and, where available, claims) and validated per protocol. Participants without an event will be censored at last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Reginald Swift, Principal Investigator — Rubix LS
Locations (1):
- Rubix LS, Lawrence, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided